CLINICAL TRIAL: NCT05395559
Title: Prevalence and Recognition of Cognitive Impairment in Hospitalized Patients: a Flash Mob Study
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Health∼Holland, Topsector Life Sciences & Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202200087
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Impairment; Dementia; Alzheimer Disease; Delirium
Keywords: Elderly; Hospitalization
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this multicenter, cross-sectional, observational flash mob study is to investigate the prevalence of cognitive impairment in hospitalized elderly aged 65 years or older, and the recognition of cognitive impairment by healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Dutch-speaking
* Hospitalized
* Age ≥ 65 years old

Exclusion Criteria:

* Unable to perform the Mini-Cog (e.g. due to visual impairment, severe hearing loss, being too ill, or otherwise unable to speak or write)
* Patients who require medical isolation
* Not willing to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient population:
  Dutch-speaking, hospitalized patients aged ≥ 65 years old.
  Healthcare professional population:
  Nurses and physicians who work at participating wards and take care of one or more participating patients.
Sampling Method: Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Percentage of hospitalized patients aged 65 years or older with cognitive impairment | Baseline
  Cognitive impairment is measured with the Mini-Cog
Percentage of hospitalized patients aged 65 years or older with cognitive impairment that has been recognized by nurses, physicians, both their nurse and physician, and either their nurse or physician | Baseline
  Cognitive impairment is measured with the Mini-Cog

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C van Munster, Prof. dr., Principal Investigator — University Medical Center Groningen, University Center for Geriatric Medicine
Locations (1):
- University Department of Geriatric Medicine, Groningen, Netherlands